CLINICAL TRIAL: NCT02345668
Title: Effectiveness of a Transdiagnostic Internet-based Treatment for Emotional Disorders vs Treatment as Usual in Specialized Care: a Randomized Controlled Trial
Brief Title: Effectiveness of a Transdiagnostic Internet-based Treatment for Emotional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Consorcio Hospitalario Provincial de Castellón (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI09
Record Dates: First submitted 2015-01-09; First posted 2015-01-26 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Depression
Keywords: Transdiagnostic Internet-based Protocol; Treatment as Usual (TAU)
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Therapeutics; Drug Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdiagnostic Internet-based Treatment (Experimental): Intervention group that carries out the Emotion Regulation Protocol and receives support by the therapist (a brief weekly two-minute phone call without clinical content and two weekly orientative text messages)
  Interventions: Behavioral: Emotion Regulation Protocol
- Treatment as Usual (Experimental): Intervention group that receives psychological and/or pharmacological treatment from a clinician of the mental health unit.
  Interventions: Drug: Treatment as Usual (Pharmacological Treatment); Behavioral: Treatment as Usual (Psychological Treatment)

INTERVENTIONS:
Behavioral: Emotion Regulation Protocol — Emotion Regulation Protocol is an Internet-based Self-administered Protocol for emotional disorders, which will allow the individual to learn and practice adaptive ways to regulate their emotions from a transdiagnostic perspective. The protocol contains the following components: present-focused emotional awareness, cognitive flexibility, emotional avoidance and emotion-driven behaviors, interoceptive and situation-based emotion exposure, psychoeducation about emotions, motivational enhancement and relapse prevention, which are organized in twelve modules: Emotional disorders and emotion regulation; Motivation for change; Understanding the role of emotions; The acceptance of emotional experiences; Practicing the acceptance; Learning to be flexible; Practicing the cognitive flexibility; The emotional avoidance; Emotion driven behaviors; Accepting and facing physical sensations; Facing emotions in the contexts in which they occur; and Relapse Prevention.
  Arms: Transdiagnostic Internet-based Treatment
Drug: Treatment as Usual (Pharmacological Treatment) — The Pharmacological Treatment provided by a psychiatrist in the mental health unit.
  Arms: Treatment as Usual
Behavioral: Treatment as Usual (Psychological Treatment) — The Psychological Treatment provided by a clinical psychologist in the mental health unit.
  Arms: Treatment as Usual

SUMMARY:
The aim of this study is to assess the efficacy of a Transdiagnostic Internet-based Protocol (Emotion Regulation Protocol) for the treatment of unipolar mood disorders (major depression and dysthimia) four anxiety disorders (Panic disorder, agoraphobia, generalized anxiety disorder and social anxiety disorder) and obsessive-compulsive disorder in comparison with Treatment as Usual in specialized care (Spanish public mental health system).

DETAILED DESCRIPTION:
Emotional disorders (ED) (anxiety and mood disorders) are among the most prevalent mental disorders, with a life prevalence of 29% and comorbidity rates that range between 40 and 80%. If they are not adequately treated the course is often chronic, and them significantly affect important functioning areas such as work and social relationships. Thus, these data strongly suggest efficacious and efficient treatments are needed in order to address this important health problem. The classification and differentiation of mental disorders carried out in manuals like the DSM and the ICD has played an important role in the emphasis placed on the research about the treatment of specific disorders; however, it has also been a problem in the dissemination of evidenced-based treatments due to the difficulties in training the clinicians in the variety of the available disorder-specific programs. In fact, less than 50% of people suffering from emotional disorders receive a psychological treatment; and this is also accounted for by its costs and time of application. As a consequence, many people decide not to search for psychological treatment. In addition, epidemiological studies have shown that at least 55% of people suffering from an anxiety disorder suffer from another anxiety disorder at the moment of the assessment, and this prevalence rate is up to 76% when different lifespan diagnoses are taken into account. This high comorbidity rate indicates that the different ED share important characteristics and it has been proposed that this overlapping is accounted for by common biological and psychological vulnerabilities that along with psychosocial stress factors leads to different manifestations of the same vulnerability, i. e., the different mood and anxiety disorders. Thus, a Transdiagnostic approach could help overcome these barriers.

Transdiagnostic approaches have implications in the treatment of psychological disorders as a number of treatment protocols have been developed based on this perspective. Clark has distinguished three perspectives in transdiagnostic cognitive-behavioral therapy: a) The transdiagnostic practice, a pragmatic perspective that includes components of various disorder-specific intervention protocols whose aim is to determine which are the active components in samples with those disorders. The contributions of Norton, Andrews and Titov, and the study: Coordinated Anxiety Learning and Management (CALM) belong to this category. b) The transdiagnostic theory, that specifies a theoretical framework which outlines the common psychological constructs that influence the maintenance of ED. For instance, the tripartite model of anxiety and depression, with positive and negative affect as relevant constructs. c) The Unified Protocol. The Barlow's team has designed a protocol, adequate for the treatment of ED which focuses on four essential aspects: to increase present-focused emotional awareness, to identify and modify emotional avoidance patterns, to promote the cognitive flexibility and to facilitate exposure to avoided situations and sensations.

Another aspect that could enhance the dissemination of evidence-based treatments as well as considerably reduce the costs is the use of the Internet. A number of sistematic reviews has shown that Internet-based treatments yield similar results when compared to face-to-face therapy. Nevertheless, most of these programs are focused on a single disorder since a few Transdiagostic Internet-based treatments have been developed and tested by means of randomized controlled trials so far. Furthermore, no studies on efficacy of Internet-based Transdiagnostic vs Treatment as usual (TAU) have been carried out in specialized care. Therefore, we have developed a Transdiagnostic Internet-based protocol treatment (Emotion Regulation Protocol) based on the Unified Protocol proposed by Barlow, that also includes components of emotion regulation and acceptance.

The aim of this study will be to test the efficacy of a Transdiagnostic Internet-based protocol (Emotion Regulation Protocol) for the treatment of emotional disorders by means of a randomized controlled trial in a sample made up of participants from specialized care of the Spanish public mental health system. The study will include two conditions: a) Transdiagnostic Internet-based treatment protocol and b) TAU. The main hypothesis is that the Transdiagnostic protocol will be more efficacious than TAU and that will obtain a good acceptance by patients and mental health professionals. We also expect the online Transdiagnostic protocol to be more efficient when compared with TAU (e. g., a significant greater number of patients which receive a psychological treatment, a significant reduction of the waiting lists and costs such as hours of clinical assistance and hours of face-to-face treatment, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18 and 70 years old.
* Meeting the DSM-IV diagnosis criteria of emotional disorder (panic disorder with or without agoraphopia, social anxiety disorder, generalized anxiety disorder, obsessive-compulsive disorder, major depression disorder and dysthimia).
* Providing written, informed consent.
* Being able to understand and read Spanish.
* Having daily acces to the Internet in their natural environment.

Exclusion Criteria:

* Being diagnosed a severe mental disorder (people with the following mental disorders will be excluded from the study: schizophrenia, bipolar disorder and personality disorders from clusters A and B).
* Being diagnosed an alcohol and/or substance dependence disorder.
* The presence of high suicidal risk.
* A medical disease or condition which prevent the participant from carry out the psychological treatment.
* Receiving another psychological treatment while the study is still ongoing.
* The increase and/or changes in the medication of participants receiving pharmacological treament during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in the Beck Depression Inventory (BDI-II) (Beck, Steer, & Brown, 1990; Sanz, Navarro, & Vázquez, 2003) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  It is one of the most widely used questionnaires to evaluate depression severity in pharmacological and psychotherapy trials. It consists of 21 items about the different symptoms characterizing major depression disorder, added together to obtain the total score, which can be a maximum of 63 points. The instrument has good internal consistency (α = 0.76 to 0.95). The Spanish version of this instrument has also shown a high internal consistency (α = 0.87) for both the general and clinical populations (α = .89) are coded from 0 to 4, added together to obtain a total score ranging from 0 to 20. The Spanish version has shown shown good internal consistency (α = 0.86), and convergent and discriminant validity.
Change in the Beck Anxiety Inventory (BAI) (Beck, & Steer, 1990; Magán, Sanz, & García-Vera, 2008) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The BAI is a 21-item self-report measure designed to assess anxiety. Each item has a 4-point Severity scale (e.g., not at all, mildly, moderately, and severely) that addresses symptoms experienced during the past week. The internal consistency of the BAI has been found to range from .85 to .94.

SECONDARY OUTCOMES:
Change in Obsessive-Compulsive Inventory (OCI-R) (Foa et al., 2002; Fullana et al., 2004) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The OCI-R is a scale made up of 18 items rated from 1 to 4 and organized in six dimensions (washing, verification, order, obsession, hoarding and mental neutralization) that assess obsessive-compulsive behaviors. The OCI-R has showed good internal consistency (α = .81 to .93), good to excellent test-retest reliability (α = .57 to .91) and good convergent validity. The internal consistency of the Spanish version of the OCI-R has been found to be good (α = .86)
Change in the Self-Reported Panic Disorder Severity Scale (PDSS-SR) (Houck, Spiegel, Shear, & Rucci, 2002) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The scale measures the severity of the panic disorder through measures of panic attack frequency, distress during the panic attacks, anticipatory anxiety, fear and agoraphobic avoidance, fear and avoidance of physical sensations, and work and social impairment. The reliability of the scale has proved to be excellent (coefficient alpha of .917) as also has done the test-retest reliability (ICC = .81).
Change in the Pen State Worry Questionnaire (PSWQ) (Meyer, Miller, Metzger, & Borkovec, 1990) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  It is a questionnaire that evaluates the worry as an incontrollable, generalized and excessive experience. The psychometric properties of the PSWQ have proved to be good, with an internal consistency ranging from .91 to .95, and a good validity and test-retest reliability.
Change in the Social Interaction Anxiety Inventory (SIAS) (Mattick y Clarke, 1998) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  This scale is made up of twenty items rated 0 to 4 that asses the anxiety experienced by the patient in social interactive situations. The scale has a good internal consistency (alpha coefficient between .88 and .94), good test-retest and discriminant reliability, as well as appropriate construct validity.

OTHER OUTCOMES:
Change in the EuroQoL-5D (Badía, 1999) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  Generic instrument of health-related quality of life. It consists of two parts: Part 1 assesses self-reported problems in each of five domains: mobility, self-care, daily activities, pain/discomfort and anxiety/depression. Each domain is divided into three levels of severity corresponding to no problems, some problems, and extreme problems Part 2 records the subject's self-assessed health on a VAS, a 10 cm vertical line on which the best and worst imaginable health states score 100 and 0, respectively.
Client Service Receipt Inventory (CSRI) (Vázquez-Barquero et al., 1997) at pre, at 3 and 12 months follow-ups. | Up to 12 months
  The CSRI is an interview that allows the clinician to collect quantitative and qualitative information about the use of health and social services, as well as information about the economic impact of the disease (e. g., time off sick from work due to the disease). The CSRI takes about 20 minutes to be administered and includes multiple choice items as well as open questions. The version utilized in this study was designed to assess the use of services in the previous twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Professor, Study Director — University Jaume I, Castellon, Spain; Azucena García-Palacios, Professor, Study Director — University Jaume I, Castellon, Spain; Francisco Traver, Study Chair — Consorcio Hospitalario Provincial de Castellón, Spain; Gonzalo Haro, Study Chair — Consorcio Hospitalario Provincial de Castellón, Spain; Ginés Llorca, Study Chair — Consorcio Hospitalario Provincial de Castellón, Spain; Alberto Gonzalez-Robles, PhD Student, Study Chair — University Jaume I, Castellon, Spain
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Titov N, Andrews G, Johnston L, Robinson E, Spence J. Transdiagnostic Internet treatment for anxiety disorders: A randomized controlled trial. Behav Res Ther. 2010 Sep;48(9):890-9. doi: 10.1016/j.brat.2010.05.014. Epub 2010 May 24. PMID 20561606
- [Background] Titov N, Dear BF, Schwencke G, Andrews G, Johnston L, Craske MG, McEvoy P. Transdiagnostic internet treatment for anxiety and depression: a randomised controlled trial. Behav Res Ther. 2011 Aug;49(8):441-52. doi: 10.1016/j.brat.2011.03.007. Epub 2011 Apr 3. PMID 21679925
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Derived] Gonzalez-Robles A, Roca P, Diaz-Garcia A, Garcia-Palacios A, Botella C. Long-term Effectiveness and Predictors of Transdiagnostic Internet-Delivered Cognitive Behavioral Therapy for Emotional Disorders in Specialized Care: Secondary Analysis of a Randomized Controlled Trial. JMIR Ment Health. 2022 Oct 31;9(10):e40268. doi: 10.2196/40268. PMID 36315227
- [Derived] Gonzalez-Robles A, Diaz-Garcia A, Garcia-Palacios A, Roca P, Ramos-Quiroga JA, Botella C. Effectiveness of a Transdiagnostic Guided Internet-Delivered Protocol for Emotional Disorders Versus Treatment as Usual in Specialized Care: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 7;22(7):e18220. doi: 10.2196/18220. PMID 32673226
- [Derived] Gonzalez-Robles A, Garcia-Palacios A, Banos R, Riera A, Llorca G, Traver F, Haro G, Palop V, Lera G, Romeu JE, Botella C. Effectiveness of a transdiagnostic internet-based protocol for the treatment of emotional disorders versus treatment as usual in specialized care: study protocol for a randomized controlled trial. Trials. 2015 Oct 31;16:488. doi: 10.1186/s13063-015-1024-3. PMID 26519046
- See also: Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es
- See also: Web site of the intervention program — http://www.psicologiaytecnologia.com